CLINICAL TRIAL: NCT05123092
Title: The Efficacy of Erector Spinae Plane Block Compared to Intrathecal Morphine for Postoperative Analgesia in Lumbar Spine Surgery Patients: A DOUBLE - BLINDED RETROSPECTIVE COMPARATIVE STUDY.
Brief Title: Erectae Spinae Block Versus Intrathecal Morphine for Postoperative Analgesis in Lumbar Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Atef Mohamed Sayed mahmoud, Principal investigator, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: M520; M520 (Other: Faculty of medicine ethical committee, Fayoum university)
Record Dates: First submitted 2021-08-13; First posted 2021-11-17 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Post-operative; Analgesia
Keywords: Ultrsound; Intrathecal; Morphine; Erectae spinae
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: The patients will be allocated in 1:1 ratio to one of the two groups:
  group erector spinae plane block (n=41), and group intrathecal morphine (n=41).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization will be done via computer-generated random numbers that will be placed in separate closed envelopes and will be opened by study investigators just after induction of general anesthesia. Neither the patients, the study investigators, the attending clinicians nor the data collectors will be aware of the allocation of groups till the study ends.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group ( ultrasound guided erectae spinae block) (Active Comparator): The same anesthesiologist who is experienced in US guided regional anesthesia will perform the block. In the group ESP, a high frequency linear US probe (HFL_50, 15_6MHz) will be placed vertically and nearly 3 cm lateral to the vertebra in the middle of the incision line. The transverse process and the overlaying erector spinae muscles (ESM) will be identified under parasagittal scanning A22 G,50 mm block needle (SONOTAP,Pajunk, Geisingen,Germany) will be inserted at a 30-40° angle in the cranial to caudal direction via an in-plane approach and advanced into the plane between the fascia of ESM and transverse process under sterile conditions. The correct needle position will be confirmed after a hydro dissection with 3 ml of isotonic saline, and then 20 ml of 0.25% bupivacaine will be injected in the interfascial plane between the rhomboideus major muscle and ESM. The local anesthetic spread will be visualized in a fascial longitudinal pattern deep to the ESM.
  Interventions: Other: Ultrasound guided lumbar erectae spinae block; Other: Intrathecal Morphine injection
- Group (Intrathecal morphine) (Active Comparator): In the group of intrathecal morphine , a lumbar puncture will be done in the lateral position via a midline approach into the level of the vertebra which exists in the middle of the incision with complete aseptic condition using 25 gauge Quincke spinal needle to give 0.3 mg of morphine (preservative free form) suspended in 0.4 ml of normal saline .
  Interventions: Other: Ultrasound guided lumbar erectae spinae block; Other: Intrathecal Morphine injection

INTERVENTIONS:
Other: Ultrasound guided lumbar erectae spinae block — One group by using ultrasound for making erectae spinae block
Other: Intrathecal Morphine injection — Injecting intrathecal morphine

SUMMARY:
The study design will be double blinded retrospective controlled comparative study.

The patients will be included in the study shoud be in the following category:

* American Society of Anesthesiologists (ASA) physical status I, II
* Age range from 18 and 70 years.

The patients will be discarded from the study shoud be in the following:

* patient refusal.
* significant renal, hepatic and cardiovascular diseases.
* Pregnancy.
* Any contraindication to regional anesthesia such as local infection or bleeding disorders.
* Chronic opioid use, history of chronic pain and cognitive disorders.
* Lumbar spine lesion revision and dural tear. Postoperative pain will be evaluated using a visual analogue scale (VAS) score as primary outcome measure.

demographic data ( Age, Weight, sex and height) , ASA classification ,mean operative times (min), time to the first rescue analgesic (min) ,intraoperative fentanyl consumption(microgram),postoperative opioid consumption ,sedation score, hemodynamics intraoperative and postoperative ( BP ,H R and oxgen saturation %) and complications as 2ry outcome measures.

DETAILED DESCRIPTION:
This study will be performed in the in the FAYOUM University hospital after the local Institutional Ethics Committee and local institutional review board approval. The study design will be double blinded retrospective controlled comparative study. A detailed informed consent will be signed by the eligible patients before recruitment and randomization.

Inclusion criteria:

* American Society of Anesthesiologists (ASA) physical status I, II patients who will be scheduled for elective lumbar surgery for one or two levels.
* Age range from 18 and 70 years.

Exclusion criteria:

* patient refusal.
* significant renal, hepatic and cardiovascular diseases.
* History of allergy to one of the study drugs.
* Pregnancy.
* Any contraindication to regional anesthesia such as local infection or bleeding disorders.
* Chronic opioid use, history of chronic pain and cognitive disorders.
* Lumbar spine lesion revision and dural tear. Randomization will be done via computer-generated random numbers that will be placed in separate closed envelopes and will be opened by study investigators just after induction of general anesthesia. Neither the patients, the study investigators, the attending clinicians nor the data collectors will be aware of the allocation of groups till the study ends.

The patients will be allocated in 1:1 ratio to one of the two groups:

group erector spinae plane block (n=41), and group intrathecal morphine (n=41).

Anesthesia procedure:

All patients will receive 150 mg ranitidine oral tablet at the night and on the morning of the operation as a premedication. Upon arrival to the operating room, standard monitors (Electrocardiogram, Pulse oximeter, Noninvasive blood pressure monitoring) will be applied and continued all over the operation. An intravenous (IV) access will be established. General anesthesia will be performed as follows: induction will be made using IV propofol (2mg/kg), atracurium (0.5mg/kg), and fentanyl

(1microgram/kg). A cuffed endotracheal tube (7-8.5) size will be placed to secure the airway .The patients will be placed in the prone position. Maintenance of anesthesia will be made using inhalational anesthesia (isoflurane) and IV atracurium according to the patients' requirements.

Block procedure:

The same anesthesiologist who is experienced in US guided regional anesthesia will perform the block. In the group ESP, a high frequency linear US probe (HFL_50, 15_6MHz) will be placed vertically and nearly 3 cm lateral to the vertebra in the middle of the incision line. The transverse process and the overlaying erector spinae muscles (ESM) will be identified under parasagittal scanning A22 G,50 mm block needle (SONOTAP,Pajunk, Geisingen,Germany) will be inserted at a 30-40° angle in the cranial to caudal direction via an in-plane approach and advanced into the plane between the fascia of ESM and transverse process under sterile conditions. The correct needle position will be confirmed after a hydro dissection with 3 ml of isotonic saline, and then 20 ml of 0.25% bupivacaine will be injected in the interfascial plane between the rhomboideus major muscle and ESM. The local anesthetic spread will be visualized in a fascial longitudinal pattern deep to the ESM. The same procedure will be performed on the contralateral side. In the group of intrathecal morphine , a lumbar puncture will be done in the lateral position via a midline approach into the level of the vertebra which exists in the middle of the incision with complete aseptic condition using 25 gauge Quincke spinal needle to give 0.3 mg of morphine (preservative free form) suspended in 0.4 ml of normal saline . Anesthesia will be discontinued at the end of the surgery and the patients will be extubated after return of spontaneous respiration .All patients will be followed for 1 hour in the post anesthesia care unit (PACU) then discharged to the ward. In the postoperative period we will give the patients multimodal analgesic regimen as following : a) paracetamol 1000 mg IV 3 times/day, b) dexketoprofen 50 mg IV once/day, c) IV pethidine 0.5mg/kg as a rescue analgesic on demand. Postoperative pain will be evaluated using a visual analogue scale (VAS 0: no pain, 10: worst pain ever) at 0 hours postoperative in PACU, then at postoperative 2., 6.,12.,24., and 48 hours at the ward by a research assistant who will be blinded to the study groups. Pethidine IV 0.5 mg/kg will be given as a rescue analgesic when the VAS score will be more than 3. The amount of pethidine consumption will be recorded between 0-12., 12-24., and 24-48 hours. The following criteria will be recorded and compared between the two groups : demographic data ( Age, Weight, sex and height) , ASA classification ,mean operative times (min), VAS scores , time to the first rescue analgesic (h) ,intraoperative fentanyl consumption(mg),postoperative opioid consumption ,sedation score, hemodynamics intraoperative and postoperative ( blood pressure ,heart rate and spo2 ) and complications. Complications include complications related to the block and the surgery (nerve damage, local anesthesia toxicity, bleeding, infection, and thromboembolism) and complications related to the general anesthesia , intrathecal morphine and IV opioids (respiratory depression , nausea and vomiting, urine retension, hypotension , bradycardia, pruritus, constipation and dizziness ).9

Primary outcome measures:

The mean VAS score (score 0 =no pain and 10 =worst pain ever ) in the two groups of the study.

Secondary outcome measures:

The secondary outcome will include the following : demographic data ( Age, Weight, height, body mass index) , ASA classification ,mean operative times (minutes), time to first rescue analgesic (minutes) ,intraoperative fentanyl consumption(micrograme),postoperative opioid consumption ,sedation score, hemodynamics intraoperative and postoperative ( blood pressure

,heart rate and spo2 ) and complications. Complications include complications related to the block and the surgery (nerve damage, local anesthesia toxicity, bleeding, infection, and thromboembolism) and complications related to the general anesthesia, intrathecal morphine and IV opioids (respiratory depression, nausea and vomiting, hypotension, bradycardia, pruritus, constipation and dizziness).

Statistical analysis and sample size estimation :

Sample size was calculated using G*power version 3.1.9.4. Previous similar studies indicated that a minimal sample size of 37 patients in each group will be needed to achieve a power level of 0.80 , alpha level of 0.05(two tailed) , will a medium effect size of 0.66 for the VAS score at 24 hours. Estimating that 10% of patients may drop out of the study due to different reasons , sample size was increased to 82 patients (41 in each group).10 Statistical analysis will be performed using SPSS version 21.0 (IBM,Armonk,NY,USA).Data are presented as mean (SD) , median [interquartile range (IQR) ], or number of patients (%) . Distribution normality will be assessed using the Kolmogorov_Smirnov test. Comparisons between groups will be made using independent t_test or Mann_Whitney U test , as appropriate. Categorical variables will be analyzed using chi_square test or Fisher exact test. A p_value less 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I, II patients who will be scheduled for elective lumbar surgery for one or two levels. • Age range from 18 and 70 years.

Exclusion Criteria:

* patient refusal.

  * significant renal, hepatic and cardiovascular diseases.
  * History of allergy to one of the study drugs.
  * Pregnancy.
  * Any contraindication to regional anesthesia such as local infection or bleeding disorders.
  * Chronic opioid use, history of chronic pain and cognitive disorders.
  * Lumbar spine lesion revision and dural tear.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
VAS score | Every 4 bours for 48 hours post operative
  The mean VAS score (score 0 =no pain and 10 =worst pain ever ) in the two groups of the study.

SECONDARY OUTCOMES:
Age | Day 1
  Age messured by (years)
Gender | Day 1
  Male or female
Height | Day 1
  Height measured by (meter)
Weight | Day 1
  Weight measured by kilogram (kg)
Body Mass Index | Day 1
  BMI measured by kilogram divided by square meter (kg/m^2)
Mean operative time | during surgery
  Sum of operative time divided by number
Intra and post-operative opoid injected | up to 48 hours
  Sum of opoid injected intra and post
Hemodynamics intra operative | Every half hour during surgery
  MABP, HR, SPO2,
Hemodynamics post-operative | Every 4 hours for 24 hours
  MABP, HR, SPO2,
Time for 1ST analgesic request | up to 48 hours
  after what time IV analgesia reequired
Complications | up to 48 hours
  complications related to the block and the surgery (nerve damage, local anesthesia toxicity, bleeding, infection, and thromboembolism) and complications related to the general anesthesia, intrathecal morphine and IV opioids (respiratory depression, nausea and vomiting, hypotension, bradycardia, pruritus, constipation and dizziness). Grades from 1
Ramsy sedation score | Every 4 hours for 24 hours
  Ramsay Sedation Scale
  1 Patient is anxious and agitated or restless, or both 3 Patient responds to commands only 4 Patient exhibits brisk response to light glabellar tap or loud auditory stimulus 5 Patient exhibits a sluggish response to light glabellar tap or loud auditory stimulus 6 Patient exhibits no response

CONTACTS AND LOCATIONS:
Locations (1):
- Atef Mohamed mahmoud, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No
Upon finishing my study and publishing an article, I will share my data upon resonable rquest.

REFERENCES:
- [Derived] Mahmoud AM, Ragab SG, Shawky MA, Masry DH, Botros JM. The Efficacy of Erector Spinae Plane Block Compared With Intrathecal Morphine in Postoperative Analgesia in Patients Undergoing Lumbar Spine Surgery: A Double-blind Prospective Comparative Study. Pain Physician. 2023 Mar;26(2):149-159. PMID 36988361